CLINICAL TRIAL: NCT02882958
Title: Validation of Software-based Fusion of Ultrasound and MRI Images of the Prostate
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Analogic Corporation (Industry)
Responsible Party: Principal Investigator, Anthony Samir, Associate Director, Ultrasound, Department of Radiology, Massachusetts General Hospital, Massachusetts General Hospital
Other Study IDs: 2015P001681
Record Dates: First submitted 2016-05-25; First posted 2016-08-30 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Radiology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators hypothesize software-based fusion/navigation will be accurate to within 3 mm of the reference standard of EM fusion. The investigators aim to evaluate the accuracy of prostate US/MRI software-based fusion/navigation technology.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for ultrasound-guided gold seeds prostate fiducial placement prior to radiotherapy

Exclusion Criteria:

* eGFR < 45 mL/min/1.73m2
* recent (within 4 weeks) kidney or liver transplant
* contraindication to prostate MRI
* patient with cardiac pacemaker

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be single center study. Subjects will be recruited from those referred to interventional radiology for ultrasound-guided prostate fiducial placement, or those planing to undergo ultrasound-guided prostate fiducial placement in radiotherapy clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prostate Volume on Actual MRI | Within one month after the fiducial placement
  A post-procedure MRI performed within one month after the fiducial placement.
Prostate Volume on US reconstruction | During the fiducial placement
  A US 3-D sweep will be performed during the fiducial placement.
Prostate Volume based on US/EM reconstruction | During the fiducial placement
  A 3-D US sweep performed during the fiducial placement and a Electromagnetic tracking data will also be acquired at the same time, and then the two series of data will be used for US/EM reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E. Samir, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Boston, Massachusetts, United States